CLINICAL TRIAL: NCT02515461
Title: Low Energy Shockwave Therapy (LE-SWT): A Novel Treatment for Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Sune Moeller Jeppesen, BSc.med, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015_LEST_KIDNEY
Record Dates: First submitted 2015-07-27; First posted 2015-08-04 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetes mellitus; Low energy shockwave therapy; Chronic Renal Insufficiency
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention: Low energy shockwave therapy (Experimental): Low energy shockwave therapy performed on both kidneys applying 3000 shocks on each kidney.
  Interventions: Device: Low energy shockwave therapy

INTERVENTIONS:
Device: Low energy shockwave therapy — Procedure: The patient lies on supine position during treatment. Kidney will be localised in line ultrasound. 3000 shockwaves at a frequency of 4 Hz are applied to each kidney per session. The kidney will be divided into three treatment areas including 1000 shockwaves applied to each treatment area.
  Patients will receive 6 sessions over 3 weeks. Treatments are carried out on day 1, day 3, day 7, day 10, day 14, and day 17 after enrollment (average time points).
  Treatment is performed using the MODULITH SLX-F2, manufactured by STORZ MEDICAL AG.

SUMMARY:
The investigators aim to investigate whether low energy shockwave therapy (LE-SWT) can preserve kidney function in diabetic patients. Participants in this study will receive LE-SWT treatment 6 times over 3 weeks. The treatment is non-invasive and has no known side effects. Previous studies have shown that LE-SWT induces angiogenesis. The investigators hypothesize that chromium-ethylenediaminetetraacetic acid (EDTA) renal clearance remains stable or increases in treated patients. Furthermore, kidney biopsy should show no signs of damage to the tissue and possibly neo-vascularization. In this project, the investigators shall also investigate LE-SWT effect on urinary markers of tubular damage and urinary nitric oxide indices. Patients' self-reported quality of life will be assessed using Short Form 36 version 2 (SF-36v2) Health Survey.

There is an 18-months follow-up on patients. Only patients between 18-65 years old with moderate chronic kidney failure from diabetes will be included.

This project is an interventional prospective study. 30 patients with moderate kidney failure will be recruited from the Department of Endocrinology, Odense University Hospital, Denmark. LE-SWT treatment will be performed in the ambulatory of Department of Urology. Patients will be hospitalized for 1 day in the Department of Nephrology when kidney biopsy is taken (two times in study period).

DETAILED DESCRIPTION:
1.0 Background

1.1 Definitions of chronic kidney disease

The Kidney Disease Outcomes Quality Initiative (K/DOQI) of the National Kidney Foundation (NKF) defines chronic kidney disease as either kidney damage or a decreased glomerular filtration rate (GFR) of less than 60 mL/min/1.73m2 for 3 or more months.

Whatever the underlying etiology, the destruction of renal mass with irreversible sclerosis and loss of nephrons leads to a progressive decline in GFR. The different stages of chronic kidney disease form a continuum in time. In 2002, K/DOQI published its classification of the stages of chronic kidney disease (CKD), as follows:

Stage 1: Kidney damage with normal or increased GFR (>90 mL/min/1.73 m2)

Stage 2: Mild reduction in GFR (60-89 mL/min/1.73 m2)

Stage 3: Moderate reduction in GFR (30-59 mL/min/1.73 m2)

Stage 4: Severe reduction in GFR (15-29 mL/min/1.73 m2)

Stage 5: Kidney failure (GFR<15 mL/min/1.73 m2)

1.2 Epidemiology

There is a rising incidence and prevalence of kidney failure with poor outcomes and high costs. The Third National Health and Examination Survey (NHANES III) estimated that the prevalence of chronic kidney disease in adults in the United States was 11% (19.2 million). The prevalence of chronic kidney disease stages 1-4 increased from 10% in 1988-1994 to 13.1% in 1999-2004. This increase is partially explained by the increase in the prevalence of diabetes and hypertension, the two most common causes of chronic kidney disease. Data from the United States Renal Data System (USRDS) show that the prevalence of chronic renal failure increased 104% between the years 1990-2001 and incidence rates have risen 30 % between 1992 and 2008.

Diabetic nephropathy is one of the most devastating complications of diabetes. It remains the leading cause of end stage renal disease (ESRD), accounting for 44% of ESRD incident cases in the United States.

1.3 Etiology

The single most important factor responsible for the increasing incidence of CKD is diabetes mellitus. Renal affection includes albuminuria, hypertension and a decline in kidney function. Blood pressure control, which is difficult to achieve in diabetics, is mandatory for long term prognosis.

1.4 Prognosis

Many patients with chronic kidney disease might progress to ESRD. The rate of the progression depends on the underlying diagnosis, on the successful implementation of secondary preventive measures and on the individual patient.

At every age, patients with ESRD on dialysis have significantly increased morbidity and mortality when compared with non-dialysis patients and individuals without kidney disease.

1.5 Treatment

The medical care of patients with chronic kidney disease usually focus on the following:

* Delaying or halting the progression of chronic kidney disease
* Treating the pathologic manifestations of chronic kidney disease

However, no treatments are available to reverse the effects of CKD.

2.0 Aim

The aim of this study is to demonstrate that Low Energy Shockwave Treatment improves or stabilizes renal function in diabetic patients - thereby potentially reducing patients' morbidity and mortality.

3.0 Hypothesis

The investigators hypothesize that Low Energy Shockwave Therapy (LE-SWT) performed on diabetic patients' kidneys with the MODULITH SLX-F2 lithotripter:

1. Increases glomerular function measured by chromium-EDTA clearance at 3, 6, and 18 months post treatment.
2. Stimulates Nitric Oxide (NO) release measured as increased levels of NO metabolites, nitrate and nitrite, and cyclic Guanosine Monophosphate (cGMP) in patients' spot urine.
3. Does not cause increased urinary levels of markers for tubular and glomerular damage, i.e. Neutrophil Gelatinase-Associated Lipocalin (NGAL) and albumin.
4. Induces angiogenesis and prevents fibrosis in kidney tissue as shown by kidney biopsy histology. Furthermore, LE-SWT protects from destruction of the glomerular basal lamina as revealed on electron microscopy.
5. Improves self-reported quality of life measured by using the Short Form 36 version 2 (SF-36v2) health survey.
6. Causes no clinical side effects

The investigators test the hypothesis in an interventional study where 30 diabetic patients with moderate chronic kidney failure are to be treated with 6 sessions of LE-SWT on kidneys over 3 weeks.

4.0 LE-SWT treatment

Lithotripter: Treatment is carried out using the MODULITH SLX-F2 with B+W or Colour Doppler Ultrasound System.

The patient lies on supine position during treatment, no need for analgesia as the energy level of the treatment is very low. Kidney will be localised in line ultrasound (no x-ray exposure).

3000 shocks at a frequency of 4 Hz are applied to each kidney, per session. The kidney will be divided into three treatment areas including 1000 shock waves applied to each treatment area. Patients will receive 2 sessions per week for 3 weeks. Shock wave therapy takes approximately 15 minutes for each kidney. Total treatment time per session is approximately 40 minutes (including 10 minutes for preparation and ultrasound localisation).

5.0 Ethical considerations

The investigators do not expect there will be any significant ethical problems with this study. Treatment with extracorporeal shockwave lithotripsy (ESWL) for kidney stones, using 10 times the energy, has been used for more than 25 years worldwide. No kidney damage has been reported after these treatments except for a hematoma if the patient was given anticoagulant treatment. Participants will be closely monitored clinically including blood and urine tests. Blood pressure will be measured after each treatment and at the specified time schedules.

Studies are planned, including chromium-EDTA clearance measurement, renography, and a kidney biopsy. The renal biopsy is done at the Department of Nephrology, Odense University Hospital, and will be performed after the department's approved instructions and, besides the risk of bleeding, is not associated with any greater risk.

Chromium-EDTA clearance is associated with a minor radiation dose. The injected tracer contains a small amount of radioactivity, which results in a radiation dose equivalent to the absorption of a standard X-ray of the lungs. According to the Health Board regulation directives, this corresponds to 0.1 mSv, or what is equal to 1/10 of background radiation. The background radiation is the radiation dose man receives annually from the environment (for example space, earth, air, drinking water and food).

Renography is also associated with a minor radiation dose. Radioactive dose is 0.7 millisievert (mSv). Load is decreased when radioactive agent is excreted in urine.

Patients have no immediate benefits of participation apart from a possible improvement of their renal function. Patients are informed both orally and in writing.

6.0 Informed consent and patient rights

Before inclusion into the project, the patient should provide written consent to participate in this clinical project after he/she has been informed both orally and in writing in a comprehensive way on the experimental important details, risks and drawbacks. The patient is also given the patient information and a copy of the signed consent form and an individual schedule for the project. Potential participants are recommended to have a third party present during the information process. They are advised that they are entitled to consideration before a final decision is taken and that the consent at any time can be withdrawn.

The patient must consent in writing. The given written and oral information and the patient's consent are confirmed by the principal investigator Sune Møller Jeppesen and patient single-handed dated signatures.

Investigator shall not undertake any study specifically required only for this clinical project before obtaining valid informed consent.

The patients' names will be kept secret. Patients will be identified for assessment and documentation of the patient number allocated to them at the start. Patients are informed of confidentiality and patient rights through participation information.

The signed informed consent forms remain with the investigator. The investigator is required to have these forms inspect on request. The investigator will keep a list containing the patients' numbers and names so that their records - if desired - could be provided at a later date. Both consent forms and the list of patient numbers must be kept for 10 years.

7.0 Perspectives of the study

The perspective of this study is to show that LE-SWT is a harmless treatment for CKD that will improve the degree of nephropathy. LE-SWT is a non-invasive and non-painful treatment and procedure is easy to perform. Currently, no treatment is available to reverse the effects of diabetic CKD and only long-term medical intervention may halt progression of the disease. Considering morbidity and mortality of affected diabetic patients and health care costs of CKD, there is a demand to explore new therapies for CKD. Given the simplicity of LE-SWT, the investigators believe there is a potential that treatment could be cost effective even for modest results although such analysis is beyond the scope of this study.

8.0 Publication policy

Results from this project are intended published in international and national medical journals. Principal investigator Sune Møller Jeppesen will be first author and Professor Lars Lund last author on the articles. Other participants will rank according to international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3: Moderate reduction in GFR in patients with diabetes mellitus (DM)

Exclusion Criteria:

* CKD stage 1, 2, 4, 5.
* Blood pressure above 140/90 mmHg
* Renography with less than 30 % differential function on one kidney
* Kidney or ureteric stone
* Obstructive uropathy
* Kidney tumor
* Chronic Urinary Tract Infection (UTI)
* Single kidney
* Bleeding disorders (coagulopathy)
* Patient on anticoagulants
* Coronary infarction during study period
* LE-SWT for other reasons and non-diabetes mellitus kidney disease
* Severe psychiatric disorder
* Kidney transplant recipient
* Pregnant or planning on becoming pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Chromium-EDTA clearance | 19 months after enrollment (average time point).
  Measurement compared to chromium-EDTA clearance prior to intervention
Histological assessment of endothelial growth in kidneys | 19 months after enrollment (average time point).
  Semi-quantitative determination of endothelium in kidney biopsy.
Nitrite, nitrate and cGMP concentrations in spot urine sample (composite outcome) | 19 months after enrollment (average time point).
  Quantitative measurements of nitric oxide indices in urine
Neutrophil Gelatinase-Associated Lipocalin (NGAL) concentration in spot urine sample. | 2 months after enrollment (average time point).
  Assessment of tubular damage in kidneys
Patient-reported quality of life | 19 monts after enrollment (average time point).
  SF-36v2 Health Survey scores
Albumin/creatinin ratio in spot urine sample | 2 months after enrollment (average time point).
  Assessment of glomerular damage in kidneys
Histological assessment of fibrosis in kidney biopsy | 19 months after enrollment (average time point).
  Semi-quantitative determination of fibrotic tissue in kidney biopsy.
Changes in glomerulus basal lamina assessed using transmission electron microscopy. | 19 months after enrollment (average time point).
  Qualitative analysis of glomerulus basal lamina using transmission electron microscopy.

SECONDARY OUTCOMES:
Chromium-EDTA clearance | 4 months and 7 months after enrollment (average time points).
  Measurement compared to chromium-EDTA clearance prior to intervention
Nitrite, nitrate and cGMP concentrations in spot urine sample (composite outcome). | Day 1, day 3, day 7, day 10, day 14, and day 17 after enrollment (average time points). Furthermore: 2 months, 4 months, 7 months, 10 months, 13 months, and 16 months after enrollment (average time points).
  Quantitative measurements of nitric oxide indices in urine
Neutrophil Gelatinase-Associated Lipocalin (NGAL) concentration in spot urine sample. | Day 1, day 3, day 7, day 10, day 14, and day 17 after enrollment (average time points).
  Assessment of tubular damage in kidneys
Albumin/creatinin ratio in spot urine sample | Day 1, day 3, day 7, day 10, day 14, and day 17 after enrollment (average time points).
  Assessment of glomerular damage in kidneys
Patient-reported quality of life | 10 months after enrollment (average time point).
  SF-36v2 Health Survey scores
24 hour blood pressure monitoring | 2 months, 4 months, 7 months, and 19 months after enrollment (average time points).
Haematoma in kidney | 2 months, 7 months, and 13 months after enrollment (average time points).
  Ultrasound investigation of kidney for haematoma and/or other structural changes. This is a qualitative investigation.
Blood creatinine concentration (estimated glomerular filtration rate) | 2 months, 4 months, 7 months, 10 months, 13 months, 16 months, and 19 months after enrollment (average time points).
  Measurement of creatinine concentration in blood sample (estimated glomerular filtration rate).
Blood urea concentration | 2 months, 4 months, 7 months, 10 months, 13 months, 16 months, and 19 months after enrollment (average time points).
  Measurement of urea concentration in blood sample.
Albumin/creatinin ratio in urine | 2 months, 4 months, 7 months, and 19 months after enrollment (average time points).
  Measurement of albumin/creatinine ratio in 24 hour urine sample
Protein concentration in urine | 2 months, 4 months, 7 months, and 19 months after enrollment (average time points).
  Measurement of protein excretion in 24 hour urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lund, Professor, Study Director — Odense University Hospital
Locations (1):
- Odense Universitetshospital, Odense, Denmark

REFERENCES:
- [Derived] Vestersager SV, Skov-Jeppesen SM, Yderstraede KB, Bistrup C, Jensen BL, Lund L. Low-intensity extracorporeal shockwave therapy in patients with diabetic kidney disease: a matched cohort study. Int Urol Nephrol. 2025 Jul;57(7):2245-2253. doi: 10.1007/s11255-025-04379-4. Epub 2025 Feb 12. PMID 39934556
- [Derived] Klomjit N, Lerman A, Lerman LO. It Comes As a Shock: Kidney Repair Using Shockwave Therapy. Hypertension. 2020 Dec;76(6):1696-1703. doi: 10.1161/HYPERTENSIONAHA.120.14595. Epub 2020 Nov 2. PMID 33131308